CLINICAL TRIAL: NCT06123494
Title: A Phase 3, Multicenter, Randomized, Open-label Study of SHR-A1811 (HER2-ADC) Compared With the Chemotherapy Treatment Chosen by the Investigators for Subjects With HER2-positive Metastatic and/or Unresectable Gastric Cancer or Gastroesophageal Junction Adenocarcinoma Who Have Progressed on or After First-line Anti-HER2 Therapy-containing Regimen
Brief Title: SHR-A1811 for Subjects With Her2-positive Gastric Cancer and Gastroesophageal Junction Adenocarcinoma After Progression on or After First-line Anti-HER2 Therapy-containing Regimen
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-308
Record Dates: First submitted 2023-11-06; First posted 2023-11-08 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: HER2-positive Advanced Gastric Cancer or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Ramucirumab; Paclitaxel; Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811 (Experimental)
  Interventions: Drug: SHR-A1811
- The investigators' choice (Active Comparator)
  Interventions: Drug: Ramucirumab / Paclitaxel/ Docetaxel/ Irinotecan

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811 6.4 mg/kg IV infusion every 3 weeks on Day 1 of each 21-day cycle
  Arms: SHR-A1811
Drug: Ramucirumab / Paclitaxel/ Docetaxel/ Irinotecan — Ramucirumab 8mg/kg，D 1,15 + Paclitaxel 80mg/m2，D1,8,15，Q4W; Paclitaxel 80mg/m2，D1,8,15，Q4W; Docetaxel 75mg/m2，D1，Q3W; Irinotecan 150mg/m2，D1，Q2W.
  Arms: The investigators' choice

SUMMARY:
This study will assess the efficacy and safety of SHR-A1811 compared with treatment chosen by the investigator in participants with HER2-positive (defined as immunohistochemistry [IHC] 3+ or IHC 2+/in situ hybridization [ISH]+) gastric or GEJ adenocarcinoma (based on [American Society of Clinical Oncology (ASCO) College of American Pathologists (CAP) guidelines who have progressed on or after a first-line anti-HER2 therapy-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, male and female;
2. Histologically or cytologically confirmed gastric or gastroesophageal junction adenocarcinoma, and unresectable locally advanced or metastatic disease
3. Prior anti-HER-2 containing treatment
4. Progression on or after first-line standard treatment (Prior neoadjuvant or adjuvant therapy can be counted as a line of therapy if the subject progressed on or within 6 months of completing neoadjuvant or adjuvant therapy);
5. Centrally confirmed HER2-positive (IHC 3+ or IHC 2+ and evidence of HER2 amplification by ISH) as classified by ASCO-CAP on a tumor biopsy
6. At least one measurable lesion according to the solid tumor response Evaluation Criteria (RECIST 1.1);
7. ECOG: 0-1;
8. Expected survival ≥12 weeks;
9. Good blood reserve and liver, kidney and coagulation function;
10. Willing to provide informed consent for study participation.

Exclusion Criteria:

1. Receive the last dose of anti-cancer therapy(including chemotherapy, radiotherapy, biological therapy, targeted therapy or immunotherapy) within 4 weeks, prior to the first dose;
2. Known allergies to monoclonal antibodies and inactive ingredients of this product, and allergies to paclitaxel, docetaxel, and irinotecan concurrently;
3. The toxicity of prior anti-tumor therapy did not recover to the level specified by CTCAE v5.0 grade evaluation ≤ Grade 1 or inclusion/exclusion criteria;
4. Clinically active central nervous system metastases;
5. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
6. Clinically significant gastrointestinal disorder by the opinion of Investigator;
7. Has a history of immunodeficiency, including a positive HIV test;
8. During the screening visits and before the first dose, unexplained fever > 38.5℃, severe infection (CTC-AE > Grade 2), and active pulmonary inflammation were indicated by screening imaging;
9. Subjects with interstitial pneumonia or with ≥ grade 3 interstitial pneumonia during prior treatment with immune checkpoint inhibitors;
10. Active hepatitis B(HBV DNA ≥ 500 IU/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA above the lower limit of detection of the analytical method);
11. Clinically significant cardiovascular disease ,such as severe/unstable angina, symptomatic congestive heart failure (NYHA ≥ Class II.), clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention, myocardial infarction within 6 months before the first dose, cerebrovascular accident (including transient ischemic attack); QTcF of 12-lead ECG was ≥470 ms; Left ventricular ejection fraction <50%; Clinically uncontrolled hypertension;
12. Had other malignancies with 5 years;
13. Pregnant or lactating women;
14. Other factors that might have led to drop out the study by the investigator opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Time from date of randomization until death (due to any cause), up to approximately 42 months
  defined as the time from date of randomization until death from any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Time from date of randomization until first objective radiographic disease progression or death (due to any cause) whichever occurs first, up to approximately 42 months
  defined as the time from date of randomization until first objective radiographic tumor progression or death from any cause, based on Investigator assessment.
Objective response rate (ORR) | From start of treatment to date of documented disease progression, up to approximately 42 months
  defined as the proportion of participants who achieve a best response of complete response (CR) or partial response (PR) using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by Investigator.
Duration of response (DoR) | Time from initial response (CR or PR) to date of documented disease progression or death (due to any cause) whichever occurs first, up to approximately 42 months
  defined time from the initial response (CR or PR) until documented tumor progression or death from any cause and based on Investigator assessment.
Disease control rate (DCR) | From start of treatment to date of documented disease progression, up to approximately 42 months
  defined as the proportion of participants who achieved CR, PR, or stable disease (SD) for a minimum of 6 weeks during study treatment, based on Investigator assessment.
AE and SAE | From time subjects signs informed consent form up to 40 days after last study dose
  Adverse events will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0.
Immunogenicity indicators of SHR-A1811: including anti-SHR-A1811 antibodies (ADA and neutralizing antibodies) | approximately 42 months
Serum concentrations of SHR-A1811 toxin-binding antibodies and free toxin SHR169265 | approximately 42 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided